CLINICAL TRIAL: NCT02402296
Title: Efficacy of β-glucan in Treatment of Localized Aggressive Periodontitis: A Short Term Double-blinded, Placebo-controlled, Randomized Clinical Trial
Brief Title: Host Modulatory Effects of β-glucan on Localized Aggressive Periodontitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Hala Helmi Hazzaa, Assistant Professor in Department of Oral Medicine, Periodontology, Diagnosis and Radiology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Al-Azhar 1-2013
Record Dates: First submitted 2015-03-06; First posted 2015-03-30 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Localized Aggressive Periodontitis
MeSH Terms: interventions — Carbohydrates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group II (test group) (Active Comparator): Included those patients who received a systemic β-1,3/1,6-D-glucan (100 mg capsule) once/ day for 40 days after scaling and root planing.
  Interventions: Drug: β-1,3/1,6-D-glucan
- Group I (control group) (Placebo Comparator): Was assigned for patients who had scaling and root planing and empty capsules filled with carbohydrates (placebo) for 40 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: β-1,3/1,6-D-glucan — 15 patients (in group II) suffering from localized aggressive periodontitis followed a strict plaque control program (within two weeks); followed by a systemic course of β-1,3/1,6-D-glucan oral supplementation for 40 days.
  Other Names: Imurril capsules 100mg
  Arms: Group II (test group)
Other: Placebo — 15 patients (in group I) suffering from localized aggressive periodontitis followed a strict plaque control program (within two weeks); followed by a systemic course of placebo capsules oral supplementation for 40 days.
  Other Names: Empty capsules filled with carbohydrates
  Arms: Group I (control group)

SUMMARY:
combining the non-surgical therapy with a well-tolerated substance that can stimulate protective immune responses like B-glucan, might effectively mount resolution pathways contributing to resolving of the chronic lesion observed in aggressive forms of periodontal disease.

DETAILED DESCRIPTION:
Aim: To investigate the efficacy of β-glucan supplementation to non-surgical periodontal therapy in localized aggressive periodontitis (LAP) patients.

Method: 30 subjects were randomly and equally assigned to receive scaling and root planing; either with placebo pills (Group I) or β-glucan (100 mg/once a day) (Group II), for 40 days. Subjects were clinically monitored on day 0 and day 91. Gingival samples were harvested from hopeless teeth sites to be investigated histologically and immunohistochemically using matrix metalloproteinase (MMP)-1 and 9 antibodies form each patient; at the same time intervals.

ELIGIBILITY:
Inclusion Criteria:

* Except for periodontitis, patients were systemically healthy as evaluated by modified Cornell medical index.
* No more than two teeth other than first molars and incisors, with probing depth (PD) ≥ 5mm, bleeding on probing (BOP), and clinical attachment level (CAL) ≥ 5mm.
* Rapid rate of attachment loss and bone destruction.
* A radiographic examination revealing an evidence of moderate to severe vertical bone loss around permanent incisors and first molar teeth.
* Every patient should have at least 20 teeth excluding third (3rd) molars, and at least an extraction-indicated tooth for a dento-periodontal affection.
* Familial aggregation.

Exclusion Criteria:

* Previous subgingival scaling and root planing, allergy to β-glucan, smoking, former smoking, pregnancy, need of antibiotic coverage for routine dental therapy, antibiotic therapy in the previous 6 months and allergy to chlorhexidine.

Ages: 20 Years to 27 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01; Primary Completion 2014-06 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hala H. Hazzaa, Professor, Principal Investigator — Al-Azhar University, Faculty of Dental and Oral Medicine (Girls Branch)

REFERENCES:
- [Background] • Prakasam A; Elavarasu SS; Natarajan RK. Antibiotics in the management of aggressive periodontitis. J Pharm Bioallied Sci. 2012; 4 (Suppl 2): S252-5. • Aurer A; Recent Advances in periodontology. Med Sci 2012; 38: 49-59. • Acar NN; Noyan Ü; Kuru L;Kadir T; Kuru B. Adjunctive systemic use of beta-glucan in the nonsurgical treatment of chronic periodontitis. Pathogenesis and treatment of periodontitis 2012; 11: 167-82. • Stashenko P; Wang CY; Riley E; Wu Y; Ostroff G; Niederman R. Reduction of infection-stimulated periapical bone resorption by the biological response modifier PGG Glucan. J Dent Res 1995; 74 (1):323-30. • Chaple CC; Srivastrava M; Hunter N; Failure of macrophage activation in destructive periodontal disease. J Pathol 1988; 186: pp.281-286.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group I (Control Group) | Group II (Test Group)
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group II (Test Group) | Group I (Control Group) | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.4 (2.37) | 25 (1.94) | 24.7 (2.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Egypt | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Assessment of Change in Clinical Attachment Level (CAL)
Description: It is the distance from the base of the pocket till the cemento-enamel junction using Williams graduated probe
Time Frame: Day 0 and day 91 post therapy
Population: A total of 30 localized aggressive periodontitis (LAP) participants were included in this study. Medical and dental histories were obtained and intraoral examinations were carried out at pre-screening visit. Patients were diagnosed to have LAP based on the clinical and radiographic findings measurements
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group I (Control Group) | Group II (Test Group)
Number analyzed (Participants) | 15 | 15
percentage of change | -14.07 (12.29) | -37.48 (17.69)

2. Secondary Outcome: Pocket Depth (PD)
Description: It is the distance from the base of the pocket till the gingival margin using Williams graduated probe
Time Frame: Day 0 and day 91 post therapy
Population: A total of 30 localized aggressive periodontitis(LAP) participants were included in this study. Medical and dental histories were obtained and intraoral examinations were carried out at pre-screening visit. Patients were diagnosed to have LAP based on the clinical and radiographic findings
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group I (Control Group) | Group II (Test Group)
Number analyzed (Participants) | 15 | 15
percentage of change | -21.84 (17.12) | -37.01 (12.31)

3. Secondary Outcome: Gingival Index (GI)
Description: Using the values of the gingival index according to (Loe & Silness, 1963); 0-no bleeding on probing
  1. delayed bleeding on probing
  2. immediate bleeding on probing
  3. spontaneous bleeding
Time Frame: Day 0 and day 91 post therapy
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group I (Control Group) | Group II (Test Group)
Number analyzed (Participants) | 15 | 15
percentage of change | -0.87 (0.83) | -75.56 (25.87)

4. Secondary Outcome: Matrix Metallo-proteinase (MMP-1&9)
Description: Their immuno-expression was assessed in the gingival samples harvested from the gingiva adjacent to hopeless teeth (planned to be extracted for dento-periodontal causes)
Time Frame: Day 0 and day 91 post therapy
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Group I (Control Group) | Group II (Test Group)
Number analyzed (Participants) | 15 | 15
percentage of change
  Percentage of change (Matrix metallo-proteinase 1) | -24.7 (4.2) | -29.5 (5.6)
  Percentage of change (Matrix metallo-proteinase 9) | -21.7 (3.9) | -36.7 (9.6)

ADVERSE EVENTS:
Arm/Group | Group I (Control Group) | Group II (Test Group)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
No limitations or caveats were reported throughout the study period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No